CLINICAL TRIAL: NCT05668377
Title: Automated Diagnostic Performance of Smartwatch ECG for Arrhythmia Detection Using the PulseAI Neural Network.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PulseAI Ltd (Industry)
Collaborators: Beacon Hospital Research Institute, Dublin, Ireland (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2022-09-29; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: PulseAI ECG Platform — Cloud-based AI-enabled ECG analysis platform

SUMMARY:
The study is to evaluate the performance of the PulseAI neural network technology at interpreting ECG data recorded using a single-lead Smartwatch (Apple Watch).

DETAILED DESCRIPTION:
Under subject consent, subjects will have a 12-lead ECG immediately followed by a smartwatch ECG. The heart rhythm and ECG interval measurements will be compared between the 12-lead ECG and smartwatch ECG.

The arrhythmias will include:

* Atrial Fibrillation/Flutter
* Tachycardia
* Bradycardia
* Premature Atrial Contractions
* Premature Ventricular Contractions

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 22 or older, able and willing to participate in the study
* Patient admitted to hospital for ablation, cardioversion, or cardiac electrophysiological exploration.
* Patient who has read the information note and has given their consent before any procedure related to the study.

Exclusion Criteria:

* Patient with a pacemaker, implantable defibrillator or cardiac resynchronisation therapy device.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants hospitalised for ablation, cardioversion or cardiac rhythm consultation.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of arrhythmia detection. | 12 months
  Evaluate the performance of arrhythmia detection by the PulseAI neural network applied to ECG data collected via the Smartwatch compared to physicians' interpretation of the 12-lead ECG.

SECONDARY OUTCOMES:
Evaluate the performance of the Apple Watch ECG interpretation Software compared to the PulseAI software | 12 months
  Evaluate the performance of the Apple Watch ECG interpretation Software compared to the PulseAI neural network
Evalaute the performance of QTc interval measurement | 12 months
  Evaluate the performance of QTc interval measurement by the PulseAI neural network applied to the Smartwatch ECG data compared to physicians' measure of the QTc interval from the 12-lead ECG.

CONTACTS AND LOCATIONS:
Overall Officials: David Burke, PhD, Principal Investigator — Beacon Hospital Research Institute, Dublin
Locations (1):
- Beacon Hospital Research Institute, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No